CLINICAL TRIAL: NCT01677156
Title: The PRESET Registry: A Registry to Evaluate Patterns of Care Associated With the Use of Corus CAD (Age/Sex/Gene Expression Score - ASGES) in Real World Clinical Care Settings
Brief Title: A Registry to Evaluate Patterns of Care Associated With the Use of Corus CAD (or ASGES) in Primary Care Settings
Acronym: PRESET
Status: Completed | Type: Observational
Sponsor: CardioDx (Industry)
Responsible Party: Sponsor
Other Study IDs: CDX_000015; PRESET (Other: CardioDx)
Record Dates: First submitted 2012-08-29; First posted 2012-08-31 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Chest Pain; Coronary Artery Disease; Cardiovascular Diseases; Coronary Heart Disease; Angina Pectoris; CAD; CVD; CHD
Keywords: ASGES; Corus CAD; Age/Sex/Gene Expression Score; Gene Expression; GES; CAD; CVD; CHD; Precision Medicine; Clinical Utility; Registry; Coronary Artery Disease; Angina Pectoris; Chest Pain; Cardiovascular Disease; Coronary Heart Disease; PRESET
MeSH Terms: conditions — Chest Pain; Coronary Artery Disease; Cardiovascular Diseases; Coronary Disease; Angina Pectoris

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Receiving Corus CAD (ASGES): Patients receiving Corus CAD (ASGES) to aid in the diagnosis of obstructive CAD
  Interventions: Diagnostic Test: CORUS CAD (ASGES)

INTERVENTIONS:
Diagnostic Test: CORUS CAD (ASGES) — Age/Sex/Gene Expression Score - ASGES

SUMMARY:
The PRESET Registry--A Registry to Evaluate Patterns of Care Associated With the Use of Corus CAD (Age/Sex/Gene Expression score - ASGES) in Real World Clinical Care Settings (PRESET)--was designed as an observational, post-market, real-world registry to evaluate patterns of care, including referrals to a cardiologist, cardiac stress testing, CT angiography, within the first month after Corus CAD (ASGES) testing.

DETAILED DESCRIPTION:
The prospective PRESET Registry (NCT01677156) enrolled stable, nonacute adult patients presenting with typical or atypical symptoms suggestive of obstructive coronary artery disease from 21 US primary care practices from August 2012 to August 2014. Demographics, clinical characteristics, and Corus CAD (Age/Sex/Gene Expression score - ASGES) results (predefined as low [ASGES <15] or elevated [ASGES >15]) were collected, as were referrals to Cardiology or further functional/anatomic cardiac testing after Corus CAD (Age/Sex/Gene Expression score - ASGES) testing. Patients were followed for 1 year post ASGES testing.

ELIGIBILITY:
Inclusion Criteria:

1. Symptoms suggestive of CAD, according to the opinion of the site registry clinician
2. Receiving Corus CAD (ASGES) to aid in the diagnosis of obstructive CAD
3. Age >= 18 years
4. Willing and able to provide written informed consent

Exclusion Criteria:

1. History of myocardial infarction (MI)
2. Current MI or acute coronary syndrome
3. Current New York Heart Association (NYHA) class III or IV congestive heart failure symptoms
4. Known/documented CAD
5. Diabetes Mellitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients presenting to their primary clinician's office with chest pain suggestive of obstructive coronary artery disease.
Sampling Method: Probability Sample
Enrollment: 713 (Actual)
Dates: Start 2012-08; Primary Completion 2014-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
To describe referral patterns for cardiac care and testing within 1 month after gene expression testing. | 1 month

SECONDARY OUTCOMES:
To describe follow up events (eg., diagnoses, non-cardiac testing, medication use, MACE) at 12 months follow up within ASGES (age, sex,gene expression score) test strata. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Zapien, MS, Study Director — CardioDx, Inc.; Mark Monane, MD, Principal Investigator — CardioDx, Inc.
Locations (13):
- United States (13):
  - Warner Family Practice, Chandler, Arizona
  - Synergy Health, Hiawassee, Georgia
  - John's Creek Primary Care, Suwanee, Georgia
  - Paul McLaughlin, MD - Family Practice, Mount Sterling, Kentucky
  - KD Health and Wellness Center, Simmesport, Louisiana
  - Doctors for Health, Omaha, Nebraska
  - TIMA Wellness, Greensboro, North Carolina
  - Dayton Internal Medicine, Dayton, Ohio
  - Northside Medical Center, Youngstown, Ohio
  - Bells Medical Clinic, Bells, Texas
  - Family Care Clinic, Bonham, Texas
  - Aldrich Internal Medicine, Dallas, Texas
  - Texas Familicare, Hurst, Texas

REFERENCES:
- [Background] Ladapo JA, Budoff M, Sharp D, Zapien M, Huang L, Maniet B, Herman L, Monane M. Clinical Utility of a Precision Medicine Test Evaluating Outpatients with Suspected Obstructive Coronary Artery Disease. Am J Med. 2017 Apr;130(4):482.e11-482.e17. doi: 10.1016/j.amjmed.2016.11.021. Epub 2016 Dec 16. PMID 27993573
- [Derived] Ladapo JA, Budoff MJ, Sharp D, Kuo JZ, Huang L, Maniet B, Herman L, Monane M. Utility of a Precision Medicine Test in Elderly Adults with Symptoms Suggestive of Coronary Artery Disease. J Am Geriatr Soc. 2018 Feb;66(2):309-315. doi: 10.1111/jgs.15215. Epub 2017 Dec 6. PMID 29210056
- See also: Am J Med. 2017 Apr;130(4):482.e11-482.e17. doi: 10.1016/j.amjmed.2016.11.021. Epub 2016 Dec 16. — https://www.ncbi.nlm.nih.gov/pubmed/?term=Clinical+Utility+of+a+Precision+Medicine+Test+Evaluating+Outpatients+with+Suspected+Obstructive+Coronary+Artery+Disease